CLINICAL TRIAL: NCT02396511
Title: Patient Treatment Protocol of TRC105 Combined With Standard-dose Bevacizumab for Two Patients With Metastatic And Refractory Choriocarcinoma
Brief Title: TRC105 Combined With Standard-dose Bevacizumab for Two Patients With Metastatic And Refractory Choriocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tracon Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 105CC201 & 105CC201B
Record Dates: First submitted 2015-03-05; First posted 2015-03-24 (Estimated); Results first posted 2019-06-11 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-05

CONDITIONS: Choriocarcinoma
MeSH Terms: conditions — Choriocarcinoma | interventions — carotuximab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TRC105 and Bevacizumab (Experimental): TRC105 weekly intravenous infusion bevacizumab every 2 weeks intravenous infusion
  Interventions: Biological: TRC105; Biological: Bevacizumab

INTERVENTIONS:
Biological: TRC105 — weekly i.v. TRC105 in combination with every 2 weeks i.v.bevacizumab, until progression or unacceptable toxicity develops
  Other Names: Chimeric Antibody (TRC105) to CD105
Biological: Bevacizumab — Every 2 weeks i.v.bevacizumab in combination with weekly i.v. TRC105, until progression or unacceptable toxicity develops

SUMMARY:
The purpose of this study is to determine whether TRC105 in combination with Bevacizumab is effective in the treatment of two patients with metastatic and refractory choriocarcinoma.

DETAILED DESCRIPTION:
Bevacizumab is a monoclonal antibody to vascular endothelial growth factor (VEGF) that inhibits angiogenesis and extends survival in patients with a wide variety of solid tumor types. TRC105 is a monoclonal antibody to CD105, an angiogenic target highly expressed on the tumor vessels and the tumor cells in choriocarcinoma. Together, these antibodies may be efficacious in metastatic and refractory choriocarcinoma, a tumor type that is highly vascular and expresses endoglin. The purpose of this study is to determine whether TRC105 in combination with Bevacizumab is effective in the treatment of two patients with metastatic and refractory choriocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness and ability to consent for self to participate in study
2. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures
3. Measurable disease by RECIST 1.1 and elevated serum β-hCG
4. Histologically proven choriocarcinoma that has progressed despite all described lines of chemotherapy for this condition

Exclusion Criteria:

1. Prior treatment with TRC105
2. Serious dose-limiting toxicity related to prior bevacizumab
3. Current treatment on another therapeutic clinical trial
4. Uncontrolled chronic hypertension defined as systolic > 140 or diastolic > 90 despite optimal therapy (initiation or adjustment of BP medication prior to study entry is allowed provided that the average of 3 BP readings at a visit prior to enrollment is < 140/90 mm Hg)
5. Symptomatic pericardial or pleural effusions
6. Uncontrolled peritoneal effusions requiring paracentesis more frequently than every 2 weeks
7. Active bleeding or pathologic condition that carries a high risk of bleeding (i.e. hereditary hemorrhagic telangiectasia)
8. Thrombolytic or anticoagulant use (except to maintain i.v. catheters) within 10 days prior to first day of study therapy
9. Cardiac dysrhythmias of NCI CTCAE grade ≥ 2 within the last 28 days
10. Known active viral or nonviral hepatitis
11. Open wounds or unhealed fractures within 28 days of starting study treatment
12. History of peptic ulcer disease or erosive gastritis within the past 6 months, unless treated for the condition and complete resolution has been documented by esophagogastroduodenoscopy (EGD) within 28 days of starting study treatment
13. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) related illness
14. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-01; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Theuer, MD, Study Director — Medical Monitor
Locations (1):
- Dana-Farber Cancer Insititue, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TRC105 and Bevacizumab
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients who enrolled in the trial who received at least a portion of a dose were included
Arm/Group | TRC105 and Bevacizumab
Number analyzed (Participants) | 2
Age, Continuous [Mean (Full Range); unit: Years] | 39.5 [37 to 42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 2
Number of Prior Regimens [Median (Full Range); unit: prior regimens] | 7 [3 to 11]

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival of Two Patients With Metastatic and Refractory Choriocarcinoma
Description: Progression Free Survival of Two Patients With Metastatic and Refractory Choriocarcinoma determined according to RECIST 1.1 including measurement of serum β- hCG. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, a measurable increase in a non-target lesion, or the appearance of new lesions. A 5 mm absolute increase is also required to guard against over calling PD when the total sum is very small.
Time Frame: Assessed every 8 weeks for up to 35 Months
Measure: Mean (Full Range); unit: Months
Arm/Group | TRC105 and Bevacizumab
Number analyzed (Participants) | 2
Months | 18 [1 to 35]

2. Primary Outcome: Objective Response Rate of Two Patients With Metastatic and Refractory Choriocarcinoma by RECIST 1.1 Including Measurement of Serum β- hCG
Description: To determine the Objective Response Rate of two patients with metastatic and refractory choriocarcinoma by RECIST 1.1 including measurement of serum β- hCG. Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) categorizes response as:
  Complete Response (CR) - Disappearance of all target lesions; Partial Response (PR) - >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Assessed every 8 weeks for up to 35 Months
Measure: Count of Participants; unit: Participants
Arm/Group | TRC105 and Bevacizumab
Number analyzed (Participants) | 2
Participants
  Response | 1
  Progression | 1

3. Secondary Outcome: Frequency and Severity of Adverse Events
Description: Adverse event frequency and severity according to CTCAE version 4.0.
Time Frame: Assessed weekly during and up to 28 days after completion of study protocol over a maximum period of 35 months.
Measure: Number; unit: Events
Arm/Group | TRC105 and Bevacizumab
Number analyzed (Participants) | 2
Events
  Total SAE's | 4
  TRC105 Related SAEs | 3

ADVERSE EVENTS:
Time Frame: Patients were followed for at least 28 days after the last dose of TRC105 study drug for adverse events, up to a maximum period of 35 months.
Arm/Group | TRC105 and Bevacizumab
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 2/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TRC105 and Bevacizumab (N=2)
Headache (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1 (1)
Malaise (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TRC105 and Bevacizumab (N=2)
Pyrexia (General disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 2 (4)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Mucosal Inflammation (General disorders) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (4)
Gingival Bleeding (Gastrointestinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Glossodynia (Gastrointestinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Gingival Pain (Gastrointestinal disorders) | 1 (4)
Chest discomfort (General disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Oral Viral Infection (Infections and infestations) | 1 (1)
Gingival Infection (Infections and infestations) | 1 (4)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (2)
Periorbital oedema (Eye disorders) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Malaise (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-17): https://cdn.clinicaltrials.gov/large-docs/11/NCT02396511/Prot_SAP_000.pdf